CLINICAL TRIAL: NCT00692861
Title: The Role of Autoimmunity in Neurologic Complications of Celiac Disease
Brief Title: Autoimmunity in Neurologic Complications of Celiac Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080153; 08-N-0153
Record Dates: First submitted 2008-06-05; First posted 2008-06-06 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2014-01-03

CONDITIONS: Ataxia
Keywords: Celiac Disease; Ataxia; Adults; Health Volunteer; HV
MeSH Terms: conditions — Ataxia; Celiac Disease

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study, done in collaboration with Cornell University in New York, will explore the potential role of the body s immune response to gluten in ataxia. Celiac disease is an autoimmune disorder that is triggered by the ingestion of wheat gluten and related proteins in genetically susceptible individuals. Some people with celiac disease also develop ataxia, which is a loss of muscle coordination, leading to imbalance. The cause of the associated ataxia is not well understood, but it is suspected to be related to the immune response towards gluten in these patients. Preliminary results indicate that antibodies in people with celiac disease can react with brain proteins, which might have a role in the associated neurologic deficits. The aim of this study is to characterize the immune response in the ataxia that is associated with celiac disease.

People 18 years of age and older with 1) ataxia and no celiac disease, 2) ataxia plus celiac disease and 3) matched healthy control subjects will be enrolled at the NIH. People with celiac disease only will be enrolled at Cornell University.

All participants have a blood sample drawn for various tests of immune function as well as genetic tests. Healthy volunteers also have a history and physical examination if they have not had one done at NIH in the past year. Some patients may require additional clinical evaluations for clinical or diagnostic reasons.

DETAILED DESCRIPTION:
Objective: To understand the role of the immune system in the neurologic complications of celiac disease (CD) or gluten sensitivity (GS).

Study population: We plan to study 15 patients with CD and ataxia, 15 patients with hereditary ataxia, and 30 healthy matched controls.

Design: Four groups of patients will be enrolled into the study. The first group will consist of patients with CD and ataxia, the second group will consist of CD patients without neurological manifestations, the third group will consist of patients with hereditary cerebellar ataxia without CD, and the final group will consist of healthy 30 race matched volunteers. The second group will not be recruited at the NIH. Standardized enzyme-linked immunosorbent assay (ELISA) techniques will used to assess the presence of synapsin I in the groups of patients. Using affinity assays, cross-reactivity of antibodies to gliadin and synapsin 1 will be evaluated. Antibody epitope mapping will be performed on those antibodies that cross-react with synapsin 1 and gliadin. HLA class II genotypic and phenotypic frequencies will be assessed and compared with the matched volunteers as an exploratory measure to look for genetic risk and protective factors in this group of patients.

Outcome measures: our outcome measures are as follows:

A. To determine whether there is an association between antibody reactivity to synapsin I and neurological deficits of CD/GS.

B. To characterize the cross-reactive antibodies in patients by determining subclass and affinity

C. To map the epitope(s) of synapsin I that are targeted in patients with cross-reactive antibodies

D. To explore HLA association in the subset of patients with CD and ataxia

ELIGIBILITY:
* INCLUSION CRITERIA:

We plan to evaluate serum and blood from patients with gluten sensitivity (including both biopsy-proven CD, and biopsy-negative cases with high anti-gliadin antibody titer) accompanied by cerebellar ataxia. Serum samples will be acquired prior to initiation of a gluten-free diet. Therefore, several inclusion criteria exist based on the study group:

INCLUSION CRITERIA FOR PATIENTS WITH CD PLUS CEREBELLAR ATAXIA:

* The patient meets criteria for CD based on the modified ESPGAN criteria
* The patient has ataxia with or without neuropathy based on clinical evaluation
* The patient is free from other neurological and psychiatric deficits
* All other known causes for ataxia have been ruled out through routine clinical evaluations
* The patient is at least 18 years old and is willing to participate in the protocol
* The patient is not taking medications that are commonly known to have immune modulating effects.
* The patient is not on a gluten free diet

INCLUSION CRITERIA FOR PATIENTS WITH HEREDITARY CEREBELLAR ATAXIA WITHOUT CD:

* The patient tested negative for serologic markers of CD (i.e. antigliadin, antireticulin, and antiendomysial antibody testing as performed under protocol 93-N-0202)
* The patient has ataxia on routine clinical examination and no other neurological or psychiatric problems
* The patient has a known autosomal dominant ataxia (i.e., SCA, DRPLA, Friedreich s ataxia, and etc).

INCLUSION CRITERIA FOR MATCHED-CONTROLS:

* They should not have CD and or ataxia based on clinical evaluation and history
* Serologic testing for antigliadin, antireticulin, and antiendomysial antibodies should reveal negative results
* They should be race and age-matched with patients with CD and the ataxia group.
* They should have no neurological or psychiatric conditions based on clinical evaluation and history
* They should not have any rheumatological or autoimmune conditions in them or in their first degree relatives.
* They should be at least 18 years of age and be able to provide consent for participation
* They should not be on any immune modulating medications.

Final diagnosis of CD will strictly follow the modified criteria of the European Society for Pediatric Gastroenterology and Nutrition (ESPGAN) and recommendations of the recently held National Institutes of Health Consensus Development Conference on Celiac Disease. Assessment and diagnosis of cerebellar ataxia will be made by magnetic resonance imaging of the brain, clinical examination and genetic testing for spinocerebellar ataxias and Friedreich s ataxia. Additional routine testing will be done if necessary to exclude other causes.

Healthy and disease control groups will be evaluated for CD and for neurological deficits. Only symptom-free, antibody-negative individuals will be recruited into these control groups. Exclusion of neurological deficits and psychiatric illness in healthy and disease control subjects will be by history and neurological examination.

EXCLUSION CRITERIA:

For all groups, if other neurological and psychiatric diagnoses are present, the individual will not qualify to participate in this study.

EXCLUSION CRITERIA FOR ALL GROUPS:

* Subject is already on a gluten-restricted diet.
* Is taking known immune modulating therapy
* Have other neurological condition (except for neuropathy) or psychiatric condition
* Not willing to have blood drawn
* Is known to have immune dysfunction
* Being pregnant leads to numerous physiological changes. It is unclear if antibody characteristics are influenced by these changes.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-06-02; Study Completion 2014-01-03

PRIMARY OUTCOMES:
Antibodies to synapsin I.

SECONDARY OUTCOMES:
Antibody characterization and HLA association

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- Cornell University, New York, New York, United States

REFERENCES:
- [Background] Alaedini A, Green PH. Narrative review: celiac disease: understanding a complex autoimmune disorder. Ann Intern Med. 2005 Feb 15;142(4):289-98. doi: 10.7326/0003-4819-142-4-200502150-00011. PMID 15710962
- [Background] Fasano A, Berti I, Gerarduzzi T, Not T, Colletti RB, Drago S, Elitsur Y, Green PH, Guandalini S, Hill ID, Pietzak M, Ventura A, Thorpe M, Kryszak D, Fornaroli F, Wasserman SS, Murray JA, Horvath K. Prevalence of celiac disease in at-risk and not-at-risk groups in the United States: a large multicenter study. Arch Intern Med. 2003 Feb 10;163(3):286-92. doi: 10.1001/archinte.163.3.286. PMID 12578508
- [Background] Tommasini A, Not T, Kiren V, Baldas V, Santon D, Trevisiol C, Berti I, Neri E, Gerarduzzi T, Bruno I, Lenhardt A, Zamuner E, Spano A, Crovella S, Martellossi S, Torre G, Sblattero D, Marzari R, Bradbury A, Tamburlini G, Ventura A. Mass screening for coeliac disease using antihuman transglutaminase antibody assay. Arch Dis Child. 2004 Jun;89(6):512-5. doi: 10.1136/adc.2003.029603. PMID 15155392